CLINICAL TRIAL: NCT05045534
Title: A Dose Block-randomized, Double-blind, Placebo Controlled, Single-/Multiple-dosing, Dose-escalation Phase 1 Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetic Characteristics of TB-840 (NASH Treatment Candidate) After Oral Administration in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of TB-840 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therasid Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TB-840-PRT-01
Record Dates: First submitted 2021-08-20; First posted 2021-09-16 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: Retinoid-related orphan receptor alpha; RORα; Agonist of RORα

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort 1 Single Dose SD1 (first dose) (Experimental): Group SD1 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 2 Single Dose SD2 (second dose) (Experimental): Group SD2 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 3 Single Dose SD3 (third dose) (Experimental): Group SD3 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 4 Single Dose SD4 (fourth dose) (Experimental): Group SD4 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 5 Single Dose SD5 (fifth dose) (Experimental): Group SD5 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 6 Single Dose SD6 (sixth dose) (Experimental): Group SD6 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 7 Single Dose SD7 (seventh dose) (Experimental): Group SD7 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 8 Single Dose SD8 (eighth dose) (Experimental): Group SD8 a first single dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 9 : Mutiple Dose MD1 (Experimental): Group MD1 a first multiple dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 10 : Mutiple Dose MD2 (Experimental): Group MD2 a first multiple dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo
- Cohort 11 : Mutiple Dose MD3 (Experimental): Group MD3 a first multiple dose of TB-840(n=6) or placebo(n=2)
  Interventions: Drug: Comparison of TB-840 treatment with Placebo

INTERVENTIONS:
Drug: Comparison of TB-840 treatment with Placebo — Single dose or Multiple Dose of TB-840 treatment
  Other Names: TB-840

SUMMARY:
TB-840(Agonist of RORα) is a candidate for NASH treatment that activates RORα(Retinoid-related orphan receptor) and its target validation for RORα and potential as a NASH treatment. This study is a dose block-randomized, double-blind, placebo-controlled, single- and multiple-ascending dose study. For each dose group, 6 subjects will be randomly assigned to the test group (TB-840) and 2 subjects will be randomly assigned to the control group (placebo). Adverse event (AE) monitoring, physical examination, vital signs, ECG, clinical laboratory test will be done for safety and tolerability assessment, and blood and urine samples will be collected for Pharmacokinetic (PK) assessment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 and ≤ 45 years at the time of screening visit
* BMI of ≥ 18.0 and ≤ 27.0 kg/m2 at the time of screening visit
* Clinically confirmed as healthy based on the medical history, physical examination, vital signs, electrocardiography (ECG), and proper laboratory tests (Subjects with values out of the normal range may participate in the study if they are deemed clinically insignificant by the investigator.)
* Agree to use medically acceptable methods of contraception by participant, his/her spouse, or partner and not to donate sperm or oocyte from the date of the first dose of the investigational product (IP) until 90 days after the last dose of the IP
* Examples of medically acceptable methods of contraception
* Females (females who use oral hormonal contraceptives and subcutaneous hormonal contraceptive implants may be excluded from the study)
* Use of an intrauterine device with a proven pregnancy failure rate
* Use of barrier method with spermicide
* Surgical sterilization (salpingectomy/tubal ligation, hysterectomy, etc.)
* Males
* Use of barrier method with spermicide
* Surgical sterilization (vasectomy, vasoligation, etc.)
* Voluntarily decided to participate in the study and provided written consent to comply with the protocol

Exclusion Criteria:

* Current or history of a clinically significant hepatic, renal, gastrointestinal, respiratory, musculoskeletal, endocrine, neuropsychiatric, hemato-oncological, or cardiovascular disease
* History of gastrointestinal diseases (e.g., Crohn's disease, ulcer, etc.) or surgery (excluding simple appendectomy or hernia repair) that may affect the absorption of the investigational products
* History of clinically significant hypersensitivity to drugs containing RORα agonist or other ingredients of the same class, or other drugs (aspirin and non-steroidal anti-inflammatory drugs, antibiotics, etc.)
* History of drug abuse or positive result from urine drug screening of drugs with concerns of drug abuse
* Subjects with any of the following results at the time of screening visit:
* Systolic blood pressure: < 90 mmHg or > 140 mmHg
* Diastolic blood pressure: < 50 mmHg or > 90 mmHg
* Heart rate: < 50 bpm or > 100 bpm
* AST: > x 1.5 ULN
* ALT: > x 1.5 ULN
* ALP: > x 1.5 ULN
* T.bil: > x 1.5 ULN
* γ-GT： > x 1.5 ULN
* Serum creatinine: > x 1.5 ULN
* Participated in another bioequivalence study or clinical study and have been exposed to an investigational product within 6 months prior to the date of the first dose of this study
* Donated whole blood within 2 months or blood components within 1 month, or received blood transfusion within 1 month prior to the date of the first dose of this study
* Use of drug-metabolizing enzyme inducer or inhibitor such as barbiturates within 1 month prior to the date of the first dose of this study
* Consumption of caffeine- or grapefruit-containing foods or beverages within 3 days prior to the date of the first dose of this study
* Use of any prescription drugs or herbal medicines within 1 month, or any over-the-counter (OTC) drugs within 1 week prior to the date of the first dose of this study (Subjects may participate in the study if such use is judged not to significantly affect the assessment of safety and pharmacokinetics by the investigator.)
* Excessive intake of caffeine, excessive intake of alcohol, or heavy smoking (caffeine > 5 units/day, alcohol > 21 units/week [1 unit = 10 mL of pure alcohol], smoking > 10 cigarettes/day)
* Unable to consume meals provided by the study site
* Prior participation in this study
* Positive result in serology tests (hepatitis B tests, human immunodeficiency virus [HIV] tests, hepatitis C tests, or syphilis tests [RPR])
* Determined inappropriate for the study by the investigator

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.03 | Up to 10 days from single ascending dose
  Incidences of treatment-emergent adverse events
Number of participants with treatment-related adverse events as assessed by CTCAE v5.03 | Up to 14 days from multiple ascending dose
  Incidences of treatment-emergent adverse events

SECONDARY OUTCOMES:
Maximum concentration of drug in plasma[Cmax] | Up to 4 days from single ascending dose
  Pharmacokinetic Profile of TB-840
Maximum concentration of drug in plasma[Cmax] | Up to 8 days from multiple ascending dose
  Pharmacokinetic Profile of TB-840
Area under the plasma drug concentration-time curve[AUC] | Up to 4 days from single ascending dose
  Pharmacokinetic Profile of TB-840
Area under the plasma drug concentration-time curve[AUC] | Up to 8 days from multiple ascending dose
  Pharmacokinetic Profile of TB-840

CONTACTS AND LOCATIONS:
Locations (1):
- Therasid Bioscience, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Hwang I, Lee SR, Kim HJ, Kim Y, Lee SW. Safety, Pharmacokinetics, and Food Effect of the RORalpha Agonist TB-840, a Novel Candidate for Metabolic Dysfunction-Associated Steatohepatitis (MASH): A Randomized First-in-Human Study in Healthy Volunteers. Life (Basel). 2025 Sep 7;15(9):1410. doi: 10.3390/life15091410. PMID 41010352